CLINICAL TRIAL: NCT07239752
Title: Influence of Maintaining Apical Patency in Post-Endodontic Pain in Molars With Necrotic Pulp and Apical Periodontitis: A Randomized Controlled Trial
Brief Title: Influence of Maintaining Apical Patency on Post-Endodontic Pain in Molars
Acronym: IMAP-Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Faiz ur rahman, post graduate trainee, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCD-Endo-Patency-001
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Periapical Periodontitis; Dental Pulp Necrosis
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patency Group (Experimental): : A #10 K-file is passively advanced 1.0 mm beyond the major apical foramen before and after each successive instrumentation size to maintain patency.
  Interventions: Procedure: Patency Group; Procedure: Standard Root Canal Instrumentation
- Non-Patency Group (Active Comparator): Participants in this group will receive standard root canal treatment where instruments are carefully confined to the root canal space and do not proceed beyond the apical foramen. All other aspects of the treatment are identical to the Experimental arm.
  Interventions: Procedure: Patency Group; Procedure: Standard Root Canal Instrumentation

INTERVENTIONS:
Procedure: Patency Group — The procedural technique of passively advancing a small endodontic file (size #10 K-file) 1 mm beyond the apical foramen before and after each larger instrument during root canal cleaning and shaping. This is done to prevent blockage of the apical portion of the canal.
Procedure: Standard Root Canal Instrumentation — Root canal instrumentation that is strictly confined to the canal space, terminating at the apical constriction (working length) and avoiding any instrumentation beyond the apical foramen.

SUMMARY:
This randomized controlled trial will investigate if maintaining apical patency-a technique where a small file is gently moved past the root's end during cleaning-affects pain after a root canal. The study will include 48 adult patients needing root canal treatment on a back molar tooth with a dead nerve and infection at the root tip. Participants will be randomly assigned to one of two groups: one where the apical patency technique is used, and one where it is not. All other treatment steps will be identical. Patients will record their pain levels on a standard scale (0-100 mm Visual Analog Scale) at 6, 12, 24, 48, and 72 hours after the procedure. The goal is to determine if this specific technique influences the intensity and duration of post-treatment pain

DETAILED DESCRIPTION:
BACKGROUND: Post-operative pain remains a significant challenge in endodontics, impacting patient satisfaction. The clinical practice of maintaining apical patency-passively keeping the apical foramen patent with a small file-is debated, with conflicting evidence on its impact on post-endodontic pain. This study aims to provide clear evidence from a robust randomized controlled trial.

OBJECTIVE: To determine the influence of maintaining apical patency on the intensity and duration of post-endodontic pain in molars with necrotic pulp and apical periodontitis.

METHODS:

Study Design: Single-center, randomized, controlled, parallel-group trial.

Setting: Department of Operative Dentistry, Saidu College of Dentistry, Swat.

Participants: 48 adult patients (aged 18-65, ASA I/II) with a single permanent molar diagnosed with necrotic pulp and symptomatic apical periodontitis. Patients with prior endodontic treatment, complex anatomy, systemic illness, pregnancy, recent analgesic use, or non-restorable teeth will be excluded.

Intervention:

Patency Group (Experimental): Following determination of working length with an electronic apex locator (verified radiographically), a pre-curved size #10 K-file will be passively advanced 1.0 mm beyond the major apical foramen before and after each successive instrumentation size.

Non-Patency Group (Active Comparator): Instrumentation will be carefully confined to the root canal space and will not proceed beyond the apical foramen.

Procedure: All participants will receive single-visit root canal treatment under local anesthesia and rubber dam isolation. Cleaning and shaping will be performed using a rotary instrument system. Irrigation will be performed with sodium hypochlorite and EDTA. Obturation will be completed with gutta-percha and sealer via a standardized technique, followed by a composite restoration.

Outcome Measure: The primary outcome is post-operative pain intensity, measured using a 100-mm Visual Analog Scale (VAS). Patients will self-record their pain levels at 6, 12, 24, 48, and 72 hours post-operatively.

Data Analysis: Data will be analyzed using SPSS Statistics v25. Descriptive statistics will summarize the data. The distribution of pain severity categories will be compared using the Chi-square test. Mean VAS scores between groups will be compared using independent samples t-tests (assuming normal distribution). A p-value of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:Adult patients aged 18-65 years.

Medically healthy, classified as American Society of Anesthesiologists (ASA) Physical Status I or II.

Presence of a single permanent molar tooth diagnosed with necrotic pulp and symptomatic apical periodontitis, and indicated for primary root canal treatment.

Patients who provide informed written consent to participate in the study. -

Exclusion Criteria:

Teeth with prior endodontic treatment or complex anatomy (e.g., calcified canals, severe curvature).

Patients with significant systemic illness (e.g., uncontrolled diabetes, immunocompromised status) or pregnancy.

History of analgesic intake within 72 hours prior to the root canal procedure.

Non-restorable teeth, teeth with severe periodontal disease (pocket depth >5mm), or teeth with root fractures.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain Intensity | 6 hours after the completion of the root canal procedure
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.
Post-operative Pain Intensity at 6 hours | 6 hours after the completion of the root canal procedure.
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.
Post-operative Pain Intensity at 12 hours | 12 hours
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.
Post-operative Pain Intensity at 48 hours | 48 hours
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.
Post-operative Pain Intensity | 12 hours after the completion of the root canal procedure
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.
Post-operative Pain Intensity | 24 hours
  Pain level measured using a 100-mm Visual Analog Scale (VAS). Patients self-report by marking a line on a 100-mm horizontal scale, where 0 mm = "no pain" and 100 mm = "worst imaginable pain". The score is the distance in mm from the left anchor.

SECONDARY OUTCOMES:
ncidence of Post-operative Pain Severity | Assessed at 6, 12, 24, 48, and 72 hours after the procedure
  The proportion of participants in each group reporting different levels of pain severity, categorized based on their VAS scores. The categories are: No Pain (VAS = 0 mm), Moderate Pain (VAS = 1-54 mm), and Severe Pain (VAS = 55-100 mm).
ncidence of Post-operative Pain Severity | Assessed at 6, 12, 24, 48, and 72 hours after the procedure. The data from all time points will be aggregated to compare the overall distribution of pain severity between groups.
  The proportion of participants in each group reporting different levels of pain severity, categorized based on their VAS scores. The categories are: No Pain (VAS = 0 mm), Moderate Pain (VAS = 1-54 mm), and Severe Pain (VAS = 55-100 mm).

IPD SHARING:
Plan to Share IPD: No